CLINICAL TRIAL: NCT05244265
Title: Mindfulness Based Stress Reduction (MBSR) for Intellectually Able Autistic Adults
Brief Title: Mindfulness Based Stress Reduction for Intellectually Able Autistic Adults
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19 pandemic hindered the group based intervention
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Tatja Hirvikoski, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MBSRautisticAdults
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Treatment Satisfaction; Participation Rate, Patient; Quality of Life; Mental Illness; Acceptance Processes; Stress, Psychological
Keywords: Autism; Adults; Intervention; MBSR
MeSH Terms: conditions — Patient Participation; Mental Disorders; Behavior; Stress, Psychological; Autistic Disorder | interventions — Mindfulness-Based Stress Reduction; Therapeutics

STUDY DESIGN:
Intervention Model Description: First study is an open feasibility study, and the second one is a RCT with two parallel group study arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Open feasibility study: no masking. RCT: during the screening, assessment of eligibility and completion of T1 (baseline), the allocation to a specific study arm is masked. After T1, all participants, care provider and investigators know which arm (group or treatment as usual) was allocated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based stress reduction (MBSR) (Experimental): The 9 session MBSR program following the manual (Kabat-Zinn, 1982).
  Interventions: Behavioral: Mindfulness-based stress reduction (MBSR)
- Treatment as usual (TAU) (Active Comparator): Participants take part in their treatment as usual in outpatient habilitation and other services.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction (MBSR) — The 8 week (plus one-day retreat) manualized MBSR program according to the manual (Kabat-Zinn, 1982).
  Arms: Mindfulness-based stress reduction (MBSR)
Behavioral: Treatment as usual (TAU) — Different interventions and support in outpatient and other services.
  Arms: Treatment as usual (TAU)

SUMMARY:
This project evaluates mindfulness based stress-reduction (MBSR), adjusted and manualized for intellectually able autistic adults. MBSR is a skills training program based on further development of cognitive behavioral therapy. The program includes eight weekly group training sessions and one full-day retreat, aiming at stress reduction and improved coping in everyday life, as well as improved mental health.

The aspiration is to make ASD-adjusted MBSR an intervention that is acceptable and accessible to individuals with autism in open clinical care. This includes considering variability in background factors such as age, comorbidity and other personal qualities and preferences.

The aim of the studies is to evaluate (1) the feasibility and (2) effectiveness of MBSR in adults (18 or over) with autism without intellectual disability, in an outpatient clinical habilitation context.

DETAILED DESCRIPTION:
Mindfulness based stress-reduction (MBSR) is a well-known skills training program used worldwide (Kabat-Zinn, 1982), with studies showing positive effects in many different conditions. The MBSR program aims at increased conscious awareness and reduced subjective stress. The intervention includes one physical meeting per week (three hours) over eight weeks' time plus one mindfulness retreat day (six hours). The intervention also incorporates meditations and other suggested tasks for participants to do by themselves in-between the group sessions. The delivery of this particular version of MBSR is adjusted to meet the needs of autistic adults, without the contents of the original MBSR program curriculum being affected. Areas that were adjusted are e.g. group size, physical environment, communication, structure, and homework.

To ensure high treatment fidelity; the MBSR teachers had teacher training following the international standard, as well as being experienced clinicians working at the habilitation services centers, with extensive knowledge about the target group. All MBSR teachers received supervision and tutoring from highly experienced certified MBSR instructor, in order to ensure that the original MBSR program was followed as closely as possible.

The studies were conducted in a clinical outpatient habilitation health care context and thus constitute an important piece in the development of support for adults with ASD. The program will have an effect on facilitating the planning and implementation of feasible and accessible interventions addressing the complex needs of this target group.

This research project consists of two studies; one open feasibility trial and one randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnose within the autism spectrum according to ICD-10, DSM-IV or DSM-5.
* Minimum ≥18 years of age.
* Adequate knowledge of the Swedish language.

Exclusion Criteria:

* Intellectual disability (IQ≤70).
* Severe mental illnesses that would hinder participation (e.g. psychosis or acute risk for suicidal behaviors).
* Drug use in the last three months.
* Poor mental health as assessed with Montgomary Åsberg Depression Rating Scale (MADRS) in combination with semi-structured interview by a clinical psychologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Study 1 (feasibility study): Treatment completion. | Immediately after intervention.
  Participants attending six or more out of the total nine occasions (eight sessions and one retreat) (≥66%) were considered completers.
Study 1 (feasibility study): Credibility as measured by the Treatment Credibility Scale (TCS: Borkovec & Nau, 1972). | Baseline compared to immediately after intervention.
  Five statements scored on a ten-point Likert scale where higher points indicate higher treatment credibility.
Study 2 (RCT): Perceived stress as measured by the Perceived stress scale (Cohen et al., 1983). | Change from baseline to immediately after the intervention.
  14 statements scored on a five-point Likert-scale (0-4) where higher points indicate higher perceived stress.

SECONDARY OUTCOMES:
Study 1 (feasibility study): Perceived stress as measured by the Perceived stress scale (Cohen et al., 1983). | Baseline compared to immediately after intervention.
  14 statements scored on a five-point Likert-scale (0-4) where higher points indicate higher perceived stress.
Study 1 (feasibility study): Symptoms of anxiety and depression as measured by Hospital anxiety and depression scale (HADS: the Swedish Lisspers et al., 1997; Zigmond & Snaith, 1983). | Baseline compared to immediately after intervention.
  14 statements scored on a four-point Likert scale from "not at all" to "very often", where higher points indicate more anxiety and depressive symptoms. In addition, sub-scales anxiety and depression were analyzed separately.
Study 1 (feasibility study): Satisfaction with life as measured by Satisfaction with life scale (SWLS: Diener et al., 1985). | Baseline compared to immediately after intervention.
  Five statements scored on a seven-point Likert-scale (1-7) where higher points indicate more satisfaction with life.
Study 1 (feasibility study): Mindfulness, assessed by Mindful attention awareness scale (MAAS: Brown & Ryan, 2003). | Baseline compared to immediately after intervention.
  15 statements and scored on a six-point Likert-scale (1-6), where higher scores indicate elevated mindful awareness.
Study 1 (feasibility study): Acceptance of the Autism diagnosis, assessed by a modified version of the Acceptance and action questionnaire (Bond et al., 2011) for ASD. | Baseline compared to immediately after intervention.
  Seven statements and scored on a seven-point Likert-scale , where higher points indicate less acceptance of the ASD diagnosis.
Study 2 (RCT): Symptoms of anxiety and depression as measured by Hospital anxiety and depression scale (HADS: the Swedish Lisspers et al., 1997; Zigmond & Snaith, 1983). | Change from baseline to immediately after the intervention.
  14 statements scored on a four-point Likert scale from "not at all" to "very often", where higher points indicate more anxiety and depressive symptoms. In addition, sub-scales anxiety and depression were analyzed separately.
Study 2 (RCT): Life satisfaction as measured by Satisfaction With Life Scale (SWLS: Diener et al., 1985). | Change from baseline to immediately after the intervention.
  Five statements scored on a seven-point (1-7) Likert-scale, where higher points indicate more satisfaction with life.
Study 2 (RCT): Five Facets Mindfulness Questionnaire | Change from baseline to immediately after the intervention.
  29 statements scored on a five-point (1-5) Likert-scale (Baer et. al., 2006). Higher points indicate higher mindful awareness.
Study 2 (RCT): Acceptance of the autism diagnosis, assessed by a modified version of the Acceptance and Action Questionnaire (AAQ: Bond et al., 2011) for ASD. | Change from baseline to immediately after the intervention.
  Seven statements scored on a seven-point (1-7) Likert-scale, where higher points indicate less acceptance of the ASD diagnosis.

OTHER OUTCOMES:
Study 1 (feasibility study and RCT): Adverse events and serious adverse events. | At any timepoint during or immediately after the intervention, i.e. not a measure that was assessed for all participants, but reported by any participant that felt he/she had experienced an adverse event.
  Events reported by participants that occured during intervention (up to 9 weeks) and may or may not be associated with participation in the intervention.